CLINICAL TRIAL: NCT06011850
Title: Comparison of the Effects of Quadratus Lumborum Block (QLB) Applied for Preemptive Analgesia on Post-operative Pain in Recipients and Donors in Renal Transplantation Surgery With Intravenous Analgesic (IVA) Group
Brief Title: Investigation of the Effects of Quadratus Lumborum Block Applied to Patients in Kidney Transplant Surgery
Status: Completed | Type: Observational
Sponsor: Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Fatma Acil,MD, Principal Investigator, Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital
Other Study IDs: 08.04.2023/484
Record Dates: First submitted 2023-08-08; First posted 2023-08-25 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Kidney Transplant Recipient; Kidney Transplant Donor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Kidney Donor QLB Group: Quadratus lumborum block (QLB) will be applied to the kidney donor in kidney transplant surgery immediately after induction of general anesthesia before the surgical incision is started.
- Kidney Donor Paracetamol Group: In kidney transplantation surgery, 1000 milligrams of Paracetamol will be administered intravenously to the kidney donor before the surgical incision is started, immediately after induction of general anesthesia.
- Kidney Recipient QLB Group: Quadratus lumborum block (QLB) will be applied to the kidney recipient in kidney transplant surgery immediately after induction of general anesthesia before the surgical incision is started.
- Kidney Recipient Paracetamol Group: In kidney transplantation surgery, 1000 milligrams of Paracetamol will be administered intravenously to the kidney recipient before the surgical incision is started, immediately after induction of general anesthesia.

SUMMARY:
This study aims to determine the most effective and long-lasting pain relief method for post-operative analgesia in kidney donor and recipient patients in kidney transplantation programme with the least invasive and least drug administration.

For this reason, it is planned to perform Quadratus lumborum plane block (QLB) in a group of patients who will be kidney donors and kidney recipients in kidney transplantation and who meet the American Society of Anesthesiologists (ASA) Physical Status Classification System 1-3 risk classification between the ages of 18-70 years, and to administer intravenous pain medication without block in another group. It is planned to include at least 84 patients in the Quadratus lumborum plan block (QLB) and Intravenous Analgesia group (IVA) without gender discrimination.

Postoperative Sedation-Agitation assessment and NRS (numeric pain scale) at 1st hour, 2nd, 6th, 12th and 24th hours, as well as possible side effects such as nausea, vomiting, shoulder pain, respiratory depression, bradycardia and hypotension, total amount of opioid analgesics consumed within 24 hours and duration of hospital stay will be observed and recorded.

DETAILED DESCRIPTION:
Plane block ultrasound-guided intra-abdominal injection into the appropriate anatomical area

* the injection will be administered immediately after general anaesthesia and intubation of the patient
* to monitor compliance with the intervention The medical files and laboratory blood tests of the patients will be examined to determine whether there are any contraindications to the intervention (patients will be excluded in case of bleeding diathesis such as intra-abdominal fluid accumulation, cystic formation, International Normalized Ratio (INR) > 2 or thrombocytopenia).

Blood pressure and heart rate values of the patient and the amount of fentanyl consumed will be recorded throughout the surgery.

The level of sedation-agitation will be evaluated during extubation at the end of surgery.

In the postoperative period, blood pressure, heart rate, pain scoring and the amount of opioid analgesic consumed will be recorded by the anaesthesiologist in the general surgery organ transplant unit and the general surgery specialist and nurses in the organ transplant service at the 1st, 2nd, 6th, 12th, and 24th hours.

The patient's satisfaction level will be evaluated and recorded 24 hours after the operation.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-70 years,
* American Society of Anesthesiologists (ASA) Physical Status Classification System I-III,
* Being a volunteer kidney recipient or volunteer donor in a kidney transplant programme under general anaesthesia

Exclusion Criteria:

* Age <18 years or > 70 years
* American Society of Anesthesiologists (ASA) Physical Status Classification System >III
* body mass index (BMI) > 35 kg/m2
* known allergy to local anaesthetics or paracetamol/tramadol
* presence of preoperative chronic pain
* presence of accumulated fluid or cystic formation in the abdomen
* presence of coagulopathy
* those who are unable to give written consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Being a kidney recipient and donor in an organ transplant program
Sampling Method: Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2023-10-03 (Actual); Primary Completion 2024-05-06 (Actual); Study Completion 2024-05-07 (Actual)

PRIMARY OUTCOMES:
Assessment of pain (NRS) level | postoperative 1st, 2nd, 6th, 12th, 24th hours
  The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable"

SECONDARY OUTCOMES:
Sedation- agitation level | Will be assessed from immediately after extubation until transfer from the recovery room to the ward.
  The Riker Sedation Agitation Scale (RSAS): identifies seven levels of sedation and agitation, which range from dangerous agitation to deep sedation, with a thorough description of patient behavior.
  Riker sedation-agitation Scale:1- Unarousable, 2 -Very Sedated, 3- Sedated, 4 Calm and Cooperative, 5 -Agitated, 6 -Very Agitated, 7 -Dangerous Agitation
Duration of first analgesic requirement | During the 24 hours postoperative period
  Time in minutes from the patient's extubation to the first analgesic requirement
Blood pressure measurement | It will be recorded 10 minutes before induction of anesthesia and every 15 minutes after intubation until the end of the operation.
  Systolic, diastolic and mean arterial pressure measurements will be recorded by invasive arterial monitoring.
Measurement of heart rate | It will be recorded 10 minutes before induction of anesthesia and every 15 minutes after intubation until the end of the operation.
  The number of heart beats per minute obtained by electrocardiographic monitoring
Amount of fentanyl consumed during the operation | During surgery
  Micrograms of fentanyl consumed during surgery
Patient satisfaction assessment | At the end of 24 hours postoperatively
  Patients' satisfaction with the quality of pain management will be assessed at 24 hours postoperatively using the following scale:
  1 = very dissatisfied; 2 = quite dissatisfied; 3 = moderate; 4 = quite satisfied; 5 = very satisfied.
Nausea-vomiting | During the 24 hours postoperative period
  Questioning about the presence/absence of nausea and/or vomiting in the postoperative period
Length of hospital stay | It is assessed for up to 12 months from the date of surgery to the date of the first documented progression or the date of death from any cause, whichever comes first
  Days of hospitalisation after the operation
Total postoperative tramadol consumption | Within 24 hours postoperatively
  milligrams

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Acil, M.D., Study Chair — Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital
Locations (1):
- Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital, Diyarbakır, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sindwani G, Sahu S, Suri A, Sureka S, Thomas M. Efficacy of ultrasound guided quadratus lumborum block as postoperative analgesia in renal transplantation recipients: A randomised double blind clinical study. Indian J Anaesth. 2020 Jul;64(7):605-610. doi: 10.4103/ija.IJA_21_20. Epub 2020 Jul 1. PMID 32792737